CLINICAL TRIAL: NCT00855764
Title: Late Phase II Study of Weekly Paclitaxel (BMS-181339) in Patients With Advanced or Recurrent Head and Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA139-388
Record Dates: First submitted 2009-03-03; First posted 2009-03-04 (Estimated); Last update posted 2010-02-04 (Estimated); Status verified 2009-10

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Paclitaxel; BMS 181339

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Paclitaxel (Experimental)
  Interventions: Drug: Paclitaxel

INTERVENTIONS:
Drug: Paclitaxel — Solution, IV, 100 mg/m2, weekly for 6 of 7 weeks, until evidence of disease progression or unacceptable side effects became apparent
  Other Names: Taxol; BMS-181339

SUMMARY:
The purpose of this study is to evaluate the efficacy and the safety of paclitaxel given weekly in patients with advanced or recurrent head and neck cancer

ELIGIBILITY:
Inclusion Criteria:

* Give written and voluntary informed consent.
* Patients with cytologically or histopathologically confirmed head and neck cancer (except for thyroid cancer)
* Patients with locally advanced head and neck cancer pretreated with surgery and/or radiotherapy (plus or minus one chemotherapy regimen) and not suitable for further radical local treatment or patients with distant metastases who may have received no or one chemotherapy regimen
* Patients must have measurable disease (lesion(s) with largest diameter of 10 mm or more)
* Patients with 4 weeks or longer interval from completion of previous therapy. (2 weeks for anti-metabolites, Biological Response Modifiers (BRM), Bisphosphonates and brain only or bone irradiation /among radiotherapy/). All reversible residual effects of previous therapy should have resolved or stabilized to the best degree, as can be reasonably expected.
* Performance Status of 0 - 2
* Patients with normal major organ functions (hematologic, hepatic and renal, etc.) and who met listed below requirements at the time of evaluation done within 2 weeks prior to the scheduled first drug administration date
* Neutrophil count: ≤ 2,000/uL
* Platelet count: ≤ 100,000/uL
* Hemoglobin: ≤ 9.0g/dL
* AST: < 100 IU/L
* ALT:< 100 IU/L
* Total bilirubin: ≤ 1.5 mg/dL
* Serum creatinine: ≤ 1.5 mg/dL
* Patients with expected survival period of at least 2 months or more from study initiation.
* Men and Women, with age range of 20 years and older to less than 75 years.

Exclusion Criteria:

* Women of childbearing potential (WOCBP) who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for up to 4 weeks after the study
* Women who are pregnant or breastfeeding
* Women with a positive pregnancy test on enrollment or prior to study drug administration
* Sexually active fertile men not using an effective method of birth control for the entire study period and for up to 8 weeks after the study
* Patients with CNS metastasis that are associated with clinical symptoms, and/or are associated with surrounding edema on CT scan or MRI, or that require concomitant therapy with steroids or anti-convulsants
* Patients with active second cancer (synchronous second cancer or the disease-free interval from the previous second primary cancer to the current cancer is less than 5 years)
* Patients with serious, uncontrolled medical illness (i.e., serious cerebrovascular disorders, uncontrolled hypertension or diabetes mellitus, severe infections or active gastric ulcer, etc.), or acute inflammatory disease, etc.
* Patients with interstitial pneumonia or pulmonary fibrosis by chest CT-scan or clinical symptoms (e.g., fever, cough, shortness of breath or dyspnea)
* Patients with body cavity fluid retention which requires treatment (or an intervention). However, those who show no re-accumulation of pleural effusion for 2 weeks or longer without use of chemotherapy drugs (BRM included) after post thoracentesis or a chest tube drainage are eligible for enrollment. In addition, those with water suction of pericardial effusion shall be ineligible for enrollment
* Patients who meet one of the following criteria;
* Either myocardial infarction or anginal attack within 6 months prior to this study participation
* Medical history of congestive heart failure
* Arrhythmia requiring treatment
* Conduction abnormality (Left bundle-branch block, Class II and above atrioventricular [AV] block)
* Patients with more than grade 1 peripheral neuropathy as graded by the NCI-CTC version 2.0 criteria
* Patients with a history of hypersensitivity due to administration of drugs containing polyoxyethylene castor oil (Cremophor EL) (e.g., cyclosporine), or hardened castor oil (e.g., vitamin preparations for injection, etc.)
* Patients with previous therapy with taxanes (e.g., paclitaxel, docetaxel)
* Patients received investigational agents within 4 weeks prior to this study participation
* Patients who are compulsorily detained for legal reasons or treatment of either a psychiatric or physical (e.g., infectious disease) illness
* Patients who don't accept use of supportive therapies, i.e., blood transfusion for anemia

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2005-10; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Response rate according to the WHO criteria | Every 4 weeks

SECONDARY OUTCOMES:
Duration of response according to the WHO criteria | Every 4 weeks
Response rate according to RECIST criteria | Every 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx